CLINICAL TRIAL: NCT04238676
Title: A Phase 1b Study Investigating the Safety, Tolerability and Efficacy of PP353 in the Treatment of Patients With Chronic Low Back Pain Associated With Vertebral Body Endplate Bone Oedema (Modic 1)
Brief Title: Persica 002 Phase 1b PP353 vs Placebo in the Treatment of Low Back Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Persica Pharmaceuticals Ltd (Industry)
Collaborators: Micron Research Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Persica 002; 2018-004488-30 (EudraCT Number); U1111-1257-2567 (Registry Identifier: WHO Universal Trial Number)
Record Dates: First submitted 2020-01-16; First posted 2020-01-23 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Chronic Low-back Pain
Keywords: Back pain; Low back pain; Lower back pain; Modic
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Intervention Model Description: Part A is open label Part B is parallel placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pharmacist and injector will not be blinded to treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PP353 (Experimental)
  Interventions: Drug: PP353
- Sham injection (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PP353 — active administered by intradiscal injection
  Arms: PP353
Other: Placebo — Sham injection
  Arms: Sham injection

SUMMARY:
A Phase 1b study to investigate the efficacy of PP353 compared to placebo in the treatment of chronic low back pain associated with bone oedema.

DETAILED DESCRIPTION:
A 2-part study. In the first part the safety, tolerability and pharmacokinetics will be assessed in up to 6 participants. In the second part, the safety, tolerability and efficacy of PP353 will be assessed in up to 40 participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years, inclusive.
* Chronic low back pain in the area associated with vertebral body endplate bone oedema (Modic 1) or vertebral body endplate bone oedema and fat (Modic 1 and 2) at a single lumbar level.
* Average LBP NRS score at screening and at Day 1 pre-randomisation ≥ 4 on chronic pain medication and ≥ 6 if not on chronic pain medication; it should be higher than the leg pain NRS score
* RMDQ-23 score ≥ 9 at screening and at Day 1 pre-randomisation.
* Current episode of chronic low back pain has lasted for ≥ 6 months at the time of randomisation.
* Bodyweight of ≥ 50 kg and ≤ 120 kg.
* Failure of standard of care therapies used by their treating physician

Exclusion Criteria:

* Any vertebra with Modic 2 only lesions which:

  1. in the opinion of the investigator, after deep palpation of the vertebral spine, is contributing to the low back pain and/or
  2. are present within 2 vertebrae from the target lumbar disc.
* The target lumbar disc has lost more than half its original anticipated height at the centre or it is < 5mm in height over the central 15 mm portion
* A clear alternative cause for back pain
* Gross facet joint degeneration or cases where the investigator believes the primary pain generator to be the facet joints
* Interventional back procedure in the 6 months prior to screening or major surgery in the 12 weeks prior to screening
* History of alcohol abuse or drugs of abuse in the past 2 years
* Any other significant illness
* Previously been treated with antimicrobial agents for their low back pain or previously received any antimicrobial intradiscal injection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 12 months
Change from baseline in Low Back Pain Numerical Rating Scale (LBP NRS) score | 12 months
  Each question will be assessed by the subject on an 11-point scale with 0 = "no pain" and 10 = "the worst possible pain you can imagine."
  The LBP NRS score throughout this protocol is defined as the average of the score of the three questions:
  1. Low back pain intensity now
  2. Worst low back pain intensity in the last 14 days
  3. Average low back pain intensity over the last 14 days

SECONDARY OUTCOMES:
Change from baseline in Low Back Pain Numerical Rating Scale (LBP NRS) score | 3, 6 & 9 months
  Each question will be assessed by the subject on an 11-point scale with 0 = "no pain" and 10 = "the worst possible pain you can imagine."
  The LBP NRS score throughout this protocol is defined as the average of the score of the three questions:
  1. Low back pain intensity now
  2. Worst low back pain intensity in the last 14 days
  3. Average low back pain intensity over the last 14 days
Change from baseline in Roland Morris Disability Questionnaire-23 score | 3, 6, 9 & 12 months
Clinically relevant improvement | 3, 6, 9 &12 months
  30 percent reduction from baseline in Roland Morris Disability Questionnaire-23 score
Change from baseline in Oswestry Disability Index | 3, 6 & 12 months
Plasma pharmacokinetics - Tdur (duration above a prescribed threshold) | 11 days
Plasma pharmacokinetics - tmax (the time at which Cmax was apparent) | 11 days
Plasma pharmacokinetics - the area under the concentration versus time curve within a dosing interval | 11 days
Plasma pharmacokinetics - Cmax (the maximum observed concentration) | 11 days
Plasma pharmacokinetics - t½ (the apparent terminal half-life) | 11 days
Plasma pharmacokinetics - CL/F (the systemic clearance calculated from plasma) | 11 days

OTHER OUTCOMES:
Change from baseline of average LBP intensity NRS daily score over a 7-day period | 3, 6, 9 & 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Duncan McHale, MBBS MRCP, Study Chair — Weatherden Ltd
Locations (10):
- Gildhøj Privathospital København, Copenhagen, Denmark
- CGM Research Trust, Christchurch, New Zealand
- Spain (2):
  - Hospital Vithas Granada, Granada
  - Hospital Universitario LA PAZ, Madrid
- United Kingdom (6):
  - Royal Preston Hospital, Preston, Lancashire
  - University Hospital Of Wales, Cardiff, Wales
  - University Hospital Coventry & Warwickshire, Coventry
  - Leeds General Infirmary, Leeds
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospital Southampton Nhs Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No